CLINICAL TRIAL: NCT02689479
Title: Evaluation of the Use of 11C-5-HTP PET to Calculate βCell Mass in Clinical Islet Transplantation (DAIT CIT-09)
Brief Title: 11C-5-HTP PET in Clinical Islet Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DAIT CIT-09
Record Dates: First submitted 2016-02-22; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Type 1 Diabetes
Keywords: Clinical Islet Transplantation; Positron Emission Tomography (PET) Computed Tomography (CT) imaging
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Magnetic Resonance Spectroscopy; Continuous Glucose Monitoring; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Positron-Emission Tomography — Dynamic scanning is performed for 60 minutes. Image acquisition is performed in 3D and reconstructed using an iterative OSEM VUEPOINT algorithm
  Other Names: Positron Emission Tomography (PET) Imaging; PET Scan
Biological: 11C-5-HTP — 150-400 MBq [11C]5-HTP (approximately 2-5 MBq/kg) is administered manually as an intravenous bolus in a intravenous catheter in the arm prior to PET imaging.
Procedure: Magnetic Resonance Imaging — Analysis will focus on adipose tissue distribution and composition in the liver.
  Other Names: MRI Scans
Procedure: Mixed-Meal Tolerance Test (MMTT)
Procedure: Continuous Glucose Monitoring System® (CGMS) — CGMS involves the subcutaneous (SC) placement of a glucose sensor connected by tubing to a pager-sized monitoring device that stores glucose data. Subjects will have the sensor placed in the clinic and wear it continuously for 72 - 84 hours (Gold) or 72-144 hours (iPro2).
Procedure: Glomerular Filtration Rate Testing
Procedure: Blood draw

SUMMARY:
In people with type I diabetes, the insulin producing cells in the pancreas have been destroyed. Presently one can only evaluate the function of the graft through laboratory tests, blood sugars and the insulin requirements. The mass of the insulin producing cells and their location are not known. The possibility to study the mass of insulin producing cells is of importance when developing new treatment regimes, in order to evaluate their efficacy on this parameter.

The researchers in this study are aiming to develop methods to measure the mass of insulin producing cells. A method (positron emission tomography, PET) previously used for the diagnosis of tumors of insulin producing cells may also be used to measure the amount of insulin producing cells in patients with type I diabetes. They plan to evaluate participants with type 1 diabetes that have undergone islet transplantation, to evaluate if PET can be used to measure the beta cell mass after islet transplantation.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be considered eligible for participation in the study:

1. Subjects who are able to provide written informed consent and comply with the procedures of the study protocol.
2. Patient that has received an islet transplant in or outside the CIT01 trial (post primary endpoint).

Exclusion Criteria:

Subjects who meet any of these criteria are not eligible for participation in the study:

1. For female subjects: Positive serum pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures at the time of PET scan +/- 2 weeks.
2. Known history of severe co-existing cardiac disease, characterized by any one of the following conditions:

   1. Recent myocardial infarction (within past 6 months).
   2. Evidence of ischemia on functional cardiac exam within the last year.
   3. Left ventricular ejection fraction <30%.
3. Persistent elevation of liver function tests at the time of study entry. Persistent Aspartate Aminotransferase (serum glutamic-oxaloacetic transaminase), Alanine Aminotransferase (serum glutamate pyruvate transaminase), Alkaline phosphatase or total bilirubin, with values >1.5 times normal upper limits will exclude a patient.
4. Treatment with any anti-diabetic medication, other than insulin, within 4 weeks of enrollment.
5. Use of any investigational agents within 4 weeks of enrollment.
6. Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The relationship between β cell mass calculated from the 11C-5-HTP PET scans and the MMTT C-peptide at 90 minutes | 8 month
  Regression methods will be used to describe the association between the beta cell mass and 90 minute c-peptide.

SECONDARY OUTCOMES:
The relationship between βcell mass calculated from the 11C-5-HTP PET and the β-score computed at the time of the PET scan | 8 month
  Regression methods will also be used to develop models to describe the relationship between the number of islets infused and the islet mass measured by PET.
The relationship between βcell mass calculated from the 11C-5-HTP PET and CPGCR computed at the time of the PET scan | 8 month
The relationship between βcell mass calculated from the 11C-5-HTP PET and number of islets transplanted (Total IEQ) | 8 month
The distribution of islets in the liver | 8 month
  Descriptive measures and scatterplots will be used to visualize the distribution of beta cells in selected regions of the liver.
The distribution of fat accumulation in the liver | 8 month
The relationship between distribution patterns in the liver and MMTT C-peptide at 90 minutes computed at the time of the PET scan | 8 month
The relationship with PET and peak C-peptide | 8 month
The relationship with PET and C-peptide AUC | 8 month
The distribution of islets in the liver related to distribution of fat accumulation in the liver as measured by MRI | 8 month
  Descriptive measures and scatterplots will be used to visualize the association between beta cells and fat deposits in the liver.
The incidence and severity of adverse events related to the PET investigation including allergic reactions | 8 month

CONTACTS AND LOCATIONS:
Overall Officials: Olle Korsgren, Principal Investigator — Uppsala University Hospital; Torbjorn Lundgren, MD, Study Chair — Karolinska University Hospital
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Uppsala University, Uppsala

REFERENCES:
- [Derived] Eriksson O, Selvaraju R, Eich T, Willny M, Brismar TB, Carlbom L, Ahlstrom H, Tufvesson G, Lundgren T, Korsgren O. Positron Emission Tomography to Assess the Outcome of Intraportal Islet Transplantation. Diabetes. 2016 Sep;65(9):2482-9. doi: 10.2337/db16-0222. Epub 2016 Jun 20. PMID 27325286
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/Pages/default.aspx